CLINICAL TRIAL: NCT02551276
Title: Role of 11 Weeks of Beta2-adrenergic Signaling and Resistance Training for Cardiac and Skeletal Muscle Hypertrophy in Men
Brief Title: Chronic Beta2-adrenergic Stimulation and Cardiac and Skeletal Muscle Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Morten Nielsen, Post.Doc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SAL-STYRKE
Record Dates: First submitted 2015-09-12; First posted 2015-09-16 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Hypertrophy in Healthy Young Men
MeSH Terms: interventions — Albuterol; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Beta2-adrenergic stimulation with salbutamol and resistance training for 10 weeks
  Interventions: Drug: Salbutamol; Other: Resistance training
- Control (Placebo Comparator): Placebo and resistance training for 10 weeks
  Interventions: Drug: Placebo; Other: Resistance training

INTERVENTIONS:
Drug: Salbutamol
  Arms: Experimental
Drug: Placebo
  Arms: Control
Other: Resistance training

SUMMARY:
Studies in animals have shown that beta2-adrenoceptor activation with selective agonists regulates protein metabolism and muscle growth in skeletal and cardiac muscle tissue. These effects may be mediated by cAMP/PKA dependent activation of several downstream sites that modulate protein synthesis and breakdown. While the role of beta2-adrenoceptor signaling is well-described in animals, it is inadequately explored in humans. The purpose of the study is thus to investigate the effect of chronic beta2-adrenergic stimulation (cAMP/PKA-signaling) on muscle hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Physical active
* Non-smokers
* Non-asthmatics
* No chronic diseases
* Informed consent

Exclusion Criteria:

* Smoker
* Allergy towards study drug

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Hypertrophy (lean body mass in Kilograms) | 2 days
  Lean body mass (kg) will be measured at two different days by Dual X-ray absorbance (DXA)

SECONDARY OUTCOMES:
Left Ventricular Hypertrophy (mass in grams) | 1 day
  Left Ventricular Mass (g) will be measured by echocardiography of the heart